**Injection Therapy in Patients with Lateral Epicondylitis** 

ID: 2018/12

**Document Date: 05/13/2018** 

**Study Protocol** 

The study was a single-blind randomized clinical trial with parallel group and allocation ratio

was 1:1. Ethical approval of the study was obtained from the Inonu University Clinical

Research Ethics Committee (No.2018/12). Volunteers meeting eligibility criteria gave

informed written consent prior to enrolment by the trial administrator. The patients who met

the inclusion criteria randomly assigned into two groups (PrT group, HA group) in a ratio of

1:1 through the stratified block randomization method. The patients and the researcher who

were responsible for the analyzing of the data were blinded to the randomization results. All

data were collected at baseline, 6 and 12 weeks. Furthermore, patients were monitored if they

had any side effects from the injection such as ecchymosis, redness, increasing pain or reduced

range of motion.

Statistical Analysis Plan

The SPSS (version23; SPSSInc., Chicago, IL, USA) was used to conduct the analysis.

Descriptive statistics were presented as mean  $\pm$  standard deviation and percentage. In the

evaluation of categorical variables, Pearson Chi-Square Test and Fisher's Final Test were used.

Suitability of variables to normal distribution were analyzed using visual (histogram and

probability graphics) and analytical methods (Shapiro-Wilk Test). Differences between the two

groups at baseline and at six and twelve weeks were tested by Independent-samples t test. Paired

t tests were used for within-group analyses. P values <0.05 were considered significant.